CLINICAL TRIAL: NCT01312051
Title: Childhood Metabolic Markers of Adult Morbidity in Blacks
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Silva Arslanian, Professor, University of Pittsburgh
Other Study IDs: R01HD027503 (NIH)
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Normal Weight; Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Protocol 1: Healthy, overweight 11 to 17 year old black and white adolescents
- Protocol 2: Healthy, normal-weight 11 to 17 year old black and white adolescents
- Protocol 3: Healthy, normal-weight 8 to 12 year old black and white adolescents
- Protocol 4: Healthy, overweight 11 to 17 year old black and white adolescents

SUMMARY:
Blacks are at increased risk for obesity, type 2 diabetes mellitus and cardiovascular disease. A common pathogenetic link among these entities is insulin resistance/hyperinsulinemia.

The specific aims of this project are: 1) to compare skeletal muscle lipid content (SMLC) in black vs white children by computed tomography (CT) scan of the mid-thigh, and assess the relationship to in vivo insulin sensitivity; 2) to test the hypothesis that free fatty acid (FFA) - induced insulin resistance is associated with larger increases in intramyocellular lipid (IMCL) in black vs white adolescents; 3) to examine if β-cell insulin secretion in prepubertal black children is more sensitive to the stimulatory effect of FFA than in whites; and 4) to test if the β-cell in black obese adolescents is more susceptible to the lipotoxic effect of FFA compared with whites. The methods to be used are: the well- established CT method as well as Magnetic Resonance Spectroscopy (1H-MRS) to assess SMLC and IMCL; intralipid infusion to elevate circulating FFA levels; the hyperinsulinemic-euglycemic clamp with stable isotopes and indirect calorimetry to measure insulin sensitivity and substrate turnover; the hyperglycemic clamp to assess insulin secretion; DEXA and whole body MRI for body composition assessments.

ELIGIBILITY:
Inclusion Criteria:

Protocols 1 & 4:

* Age 11-17 years
* Male or Female
* Healthy
* Obese, BMI ≥ 95 percentile
* Pubertal/Tanner Stage II-V
* African American or White American, based on self identity with no admixture for 3 generations

Protocol 2:

* Age 11-17 years
* Male or Female
* Healthy
* Normal Weight, BMI 10- 95 percentile
* Pubertal/Tanner Stage II-V
* African American or White American, based on self-identity with no admixture for 3 generations

Protocol 3:

* Age 8-12 years
* Male or Female
* Healthy
* Normal Weight, BMI 10-95 percentile
* Prepubertal/Tanner Stage I
* African American or White American, based on self-identity with no admixture for 3 generations

Exclusion Criteria:

* Medications which interfere with metabolism
* Hemocue < 12 gm/dl in pubertal subjects and <11gm/dl in prepubertal subjects
* Positive serum pregnancy test
* Recent significant weight change or dieting
* Presence of disease (i.e.diabetes, hypothyroidism, genetic dyslipidemia, etc)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy black and white volunteers who are 8 to 17 years of age
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2004-07; Primary Completion 2011-09-20 (Actual); Study Completion 2011-09-20 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle lipid content, insulin sensitivity and insulin secretion | Assessments at 2 timepoints occur within a 2 to 3 week period

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States